CLINICAL TRIAL: NCT00531414
Title: Inspiratory Flow and VOlumes in Asthmatic and Healthy Individuals Using the Osmohaler
Brief Title: Inspiratory Flow Using the Osmohaler
Status: Completed | Type: Observational
Sponsor: Syntara (Industry)
Other Study IDs: DPM-OSM-401
Record Dates: First submitted 2007-09-16; First posted 2007-09-18 (Estimated); Last update posted 2008-04-10 (Estimated); Status verified 2008-04

CONDITIONS: Asthma
Keywords: Asthmatic; healthy
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The OsmohalerTM is a registered device in Australia. It is used to deliver a dry powder a commercial preparation of mannitol registered as AridolTM to test if a person has irritable airways such as active asthma.

The overseas regulatory authorities need to know that people of all ages can achieve an adequate inspiratory flow through this device during a controlled deep inspiration. Adequate flow is generally regarded as greater than 30 litres per minute in children and 60 litres per minute in adults. The OsmohalerTM is a device with low resistance and is already in use in Australia to deliver mannitol. However there is a need to document inspiratory flows through the device during a controlled deep inspiration. The protocol requires subjects to perform a controlled deep inspiration from the device on three or five occasions. No substance will be inhaled.

ELIGIBILITY:
Inclusion Criteria:

* has asthma or is healthy
* aged 6 to 69 years inclusive
* FEV1 >/= 70% predicted

Exclusion Criteria:

* has condition contraindicating performance of spirometrt

Ages: 6 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2007-11; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Anderson, Principal Investigator — Royal Prince Alfred Hospital, Sydney, Australia